CLINICAL TRIAL: NCT05399485
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Rimegepant for Migraine Prevention in Japanese Subjects
Brief Title: Efficacy and Safety Study of Rimegepant for Migraine Prevention in Japanese Subjects (Japan Only)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BHV3000-309; C4951021 (Other: Alias Study Number)
Record Dates: First submitted 2022-05-27; First posted 2022-06-01 (Actual); Results first posted 2025-07-14 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Migraine
Keywords: Migraine; Headache; Migraine Prevention
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — rimegepant sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Rimegepant (Experimental): Randomization Phase: one 75 mg rimegepant (BHV3000) oral disintegration tablet every other day until Week 12
  Interventions: Drug: Rimegepant
- Placebo (Placebo Comparator): Randomization Phase: one matching placebo every other day until week 12
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rimegepant — Randomization Phase: Rimegepant (BHV3000) 75 mg orally disintegrating tablet every other day until Week 12
  Other Names: BHV3000
  Arms: Rimegepant
Drug: Placebo — Randomization Phase: Placebo tablet to match Rimegepant every other day until Week 12
  Arms: Placebo

SUMMARY:
This study is being conducted to evaluate the efficacy, safety, and tolerability of rimegepant in Japanese subjects for the prevention of migraine.

ELIGIBILITY:
Inclusion Criteria:

Subject has at least 1 year history of migraine (with or without aura) consistent with a diagnosis according to the International Classification of Headache Disorders, 3rd Edition, including the following:

1. Age of onset of migraines prior to 50 years of age.
2. Migraine attacks, on average, lasting 4 to 72 hours if untreated.
3. Per subject report, 4 to18 migraine attacks of moderate or severe intensity per month within the last 3 months prior to the Screening Visit (month is defined as 4 weeks for the purpose of this protocol).
4. 4 or more migraine days during Observation Period.
5. Not more than 18 headache days during the Observation Period.
6. Ability to distinguish migraine attacks from tension/cluster headaches.
7. Subjects on prophylactic migraine medication are permitted to remain on therapy if the dose has been stable for at least 3 months (12 weeks) prior to the Observation Period, and the dose is not expected to change during the course of the study.
8. Subjects with contraindications for use of triptans may be included provided they meet all other study entry criteria.

Exclusion Criteria:

1. Subject has a history of migraine with brainstem aura (basilar migraine), hemiplegic migraine or retinal migraine.
2. Subjects with headaches occurring 19 or more days per month (migraine or non-migraine) in any of the 3 months prior to the Screening Visit.
3. History of systemic use of analgesics (e.g. nonsteroidal anti-inflammatory drugs [NSAIDs] or acetaminophen) on ≥ 15 days per month during the 3 months (12 weeks) prior to the Screening Visit.
4. Subject with a history of HIV disease.
5. Subject history with current evidence of uncontrolled, unstable or recently diagnosed cardiovascular disease, such as ischemic heart disease, coronary artery vasospasm, and cerebral ischemia. subjects with Myocardial Infarction (MI), Acute Coronary Syndrome (ACS),Percutaneous Coronary Intervention (PCI), cardiac surgery, stroke or transient ischemic attack (TIA) during the 6 months prior to screening.
6. Uncontrolled hypertension, or uncontrolled diabetes (however subjects can be included who have stable hypertension and/or diabetes for 3 months prior to screening).
7. Subject with other pain syndromes, psychiatric conditions, dementia, or significant neurological disorders (other than migraine) that, in the Investigator's opinion, might interfere with study assessments.
8. Subject has a history of gastric, or small intestinal surgery (including Gastric Bypass, Gastric Banding, Gastric Sleeve, Gastric Balloon, etc.), or has disease that causes malabsorption.
9. The subject has a history or current evidence of any unstable medical conditions (e.g., history of congenital heart disease or arrhythmia, known or suspected infection, hepatitis B or C, or cancer) that, in the investigator's opinion, would expose them to undue risk of a significant adverse event (AE) or interfere with assessments of safety or efficacy during the course of the trial.
10. History of, treatment for, or evidence of, alcohol or drug abuse within the past 12 months or subjects who have met DSM-V criteria for any significant substance use disorder within the past 12 months from the date of the screening visit.
11. Participation in any other investigational clinical trial while participating in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 496 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (44):
- Japan (44):
  - Medical Corporation Seikokai Takanoko Hospital, Matsuyama, Ehime
  - Jinnouchi Neurosurgical Clinic, Kasuga-shi, Fukuoka
  - Ikeda Neurosurgical Clinic, Kasuga-shi, Fukuoka
  - SUBARU Health Insurance Society Ota Memorial Hospital, Ota-shi, Gunma
  - Doi Clinic Internal Medicine/Neurology, Hiroshima, Hiroshima
  - Japanese Red Cross Asahikawa Hospital, Asahikawa-shi, Hokkaido
  - Nakamura Memorial Hospital, Chūōku, Hokkaido
  - Higashi Sapporo Neurology and Neurosurgery Clinic, Sapporo, Hokkaido
  - Konan Medical Center, Higashinada-ku, Hyōgo
  - Nishinomiya Munic. Ctr. Hosp., Nishinomiya-shi, Hyōgo
  - Mito Kyodo General Hospital, Mito, Ibaraki
  - Kijima Neurosurgery Clinic, Kahoku-gun, Ishikawa-ken
  - Iwate Medical University Uchimaru Medical Center, Morioka, Iwate
  - Atsuchi Neurosurgery Hospital, Kagoshima, Kagoshima-ken
  - Tanaka Neurosurgical Clinic, Kagoshima, Kagoshima-ken
  - St. Marianna Univ. Hospital, Kawasaki-shi, Kanagawa
  - Fujitsu Clinic, Nakahara, Kanagawa
  - Atago Hospital, Kochi, Kochi
  - Umenotsuji Clinic, Kochi, Kochi
  - Saiseikai Kumamoto Hospital, Kumamoto, Kumamoto
  - Tatsuoka Neurology Clinic, Kyoto, Kyoto
  - Sendai Headache and Neurology Clinic, Medical Corporation, Sendai, Miyagi
  - Ooba Clinic for Neurosurgery & Headache, Ōita, Oita Prefecture
  - Makabe Clinic, Okayama, Okayama-ken
  - Okayama City General Medical Center Okayama City Hospital, Okayama, Okayama-ken
  - Medical Research Institute KITANO HOSPITAL, PIIF Tazuke-kofukai, Osaka, Osaka
  - Tominaga Clinic, Osaka, Osaka
  - Kindai University Hospital, Osakasayama-shi, Osaka
  - Takase Intern. Med. Clinic, Toyonaka-shi, Osaka
  - Saitama Medical University Hospital, Iruma-gun, Saitama
  - Saitama Neuropsychiatric Institute, Saitama-shi, Saitama
  - Japanese Red Cross Shizuoka Hospital, Shizuoka, Shizuoka
  - Dokkyo Medical Univ. Hosp., Shimotsuga-gun, Tochigi
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Tokai univ. hachioji hosp., Hachioji-shi, Tokyo
  - Shinagawa Strings Clinic, Minato-ku, Tokyo
  - Kitasato University Kitasato Institute Hospital, Minato-ku, Tokyo
  - USUDA CLINIC for internal medicine, Setagaya-ku, Tokyo
  - Fukuuchi Pain Clinic, Shinjuku-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Nishiogi Pain Clinic, Suginami-ku, Tokyo
  - Sakura Neuro Clinic, Toyama, Toyama
  - Nagamitsu Clinic, Hofu-shi, Yamaguchi
  - Nagaseki Headache Clinic, Kai-shi, Yamanashi

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Kitamura S, Matsumori Y, Yamamoto T, Ishikawa T, Hoshino Y, Yoshimatsu H, Thiry A, Arakawa A, Croop R, Fullerton T, Sakai F, Takeshima T. Efficacy and safety of rimegepant for the preventive treatment of migraine in Japan: A double-blind, randomized controlled trial. Headache. 2025 Sep;65(8):1403-1412. doi: 10.1111/head.14995. Epub 2025 Jun 20. PMID 40542538
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=BHV3000-309

RESULTS

PARTICIPANT FLOW:
Groups:
- Rimegepant: Participants received Rimegepant (RMG) at a dose of 75 mg, orally as an orally disintegrating tablets (ODT), once every other day (EOD) for 12 weeks in the double-blind treatment (DBT) period. Eligible participants continued to receive RMG in a similar way from Week 12 to Week 52 (40 weeks) in the OLE period.
- Placebo: Participants received placebo, orally as an ODT, once EOD for 12 weeks in the DBT period. Eligible participants continued to received Rimegepant at a dose of 75 mg, orally as an ODT from Week 12 to Week 52 (40 weeks) in the OLE period.
Period: DBT Phase
Arm/Group | Rimegepant | Placebo
Started | 247 | 249
Completed | 233 | 238
Not Completed | 14 | 11
Not completed — Other | 6 | 5
Not completed — Protocol-specified withdrawal criterion met | 1 | 1
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Protocol Violation | 2 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Adverse Event | 2 | 1
Period: OLE Phase
Arm/Group | Rimegepant | Placebo
Started | 227 (Period is for OLE phase.) | 231 (Period is for OLE phase.)
Completed | 204 | 215
Not Completed | 23 | 16
Not completed — Protocol deviation | 1 | 0
Not completed — Other | 5 | 5
Not completed — Withdrawal by Subject | 12 | 7
Not completed — Pregnancy | 0 | 2
Not completed — Physician Decision | 3 | 0
Not completed — Adverse Event | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Rimegepant: Participants received Rimegepant at a dose of 75 mg, orally as an ODT, once EOD for 12 weeks in the DBT period. Eligible participants continued to receive RMG in a similar way from Week 12 to Week 52 (40 weeks) in the OLE period.
- Placebo: Participants received placebo, orally as an ODT, once EOD for 12 weeks in the DBT period. Eligible participants continued to receive Rimegepant at a dose of 75 mg, orally as an ODT from Week 12 to Week 52 (40 weeks) in the OLE period.
- Total: Total of all reporting groups
Arm/Group | Rimegepant | Placebo | Total
Number analyzed (Participants) | 247 | 249 | 496
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.9 (9.52) | 43.1 (10.68) | 44.0 (10.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 225 | 221 | 446
  Male | 22 | 28 | 50
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Number of Migraine Days Per Month From Week 9 to 12 of the Double-Blind Treatment (DBT) Phase
Description: Migraine day: 1) day of electronic diary (eDiary) efficacy data with a qualified migraine headache, defined as: Headache lasted for >= 30 minutes and had 2 or more of following pain features: Unilateral and pulsating, moderate or severe pain intensity, worsen or avoid physical activity with one or more of the following associated symptoms: nausea, vomiting, both photophobia and phonophobia or 2) Acute migraine-specific medication day as eDiary efficacy data with a "yes" response to either of the 2 questions about taking triptan or ergotamine to treat headache or non-scheduled OL Rimegepant dosing day. The number of migraine days per month were prorated to 28 days and derived for month (i.e., 4-week interval) in on-DBT efficacy analysis period as follows: 28*(total number of migraine days in month [Week 9 to 12])/ (total number of efficacy data days in month [Week 9 to 12]).
Time Frame: Baseline, Week 9 to Week 12 of the DBT phase
Population: DBT migraine analysis set included participants in the DBT efficacy analysis set with >= 14 days of eDiary data (not necessarily consecutive) in both the observation period (OP) and >= 1 month (4-week interval) during the DBT Phase.
Measure: Least Squares Mean (95% Confidence Interval); unit: Days/month
Groups:
- Rimegepant: Participants received Rimegepant at a dose of 75 mg orally as an ODT, once EOD for 12 weeks in the DBT period.
- Placebo: Participants received placebo, orally as an ODT, once EOD for 12 weeks in the DBT period.
Arm/Group | Rimegepant | Placebo
Number analyzed (Participants) | 240 | 244
Days/month | -2.4 [-2.93 to -1.96] | -1.4 [-1.87 to -0.91]
Statistical Analysis 1: Comparison: Rimegepant vs Placebo; Linear mixed effects model with repeated measures with number of total migraine days per month in the OP as a covariate, treatment group, randomization stratum (stable prophylactic migraine medication use throughout randomization), month, and month-by treatment group interaction as fixed effects; Test type: Superiority; p = 0.0021, Mixed Models Analysis; [Difference in Least square (LS) Mean] = -1.1, 95% CI 2-sided [-1.73 to -0.38]

2. Secondary Outcome: Percentage of Participants With at Least 50% Reduction From Baseline in the Mean Number of Moderate to Severe Migraine Days Per Month in the Last 4 Weeks (Weeks 9 to 12) of the DBT Phase
Description: Percentage of participants with >= 50% reduction, from baseline in mean number of pain intensity (moderate or severe) in each month of DBT phase are included in this outcome measure. Migraine days per month are assessed as "migraine days per 4 weeks" to correspond with the 4-week visit schedule. Migraine days per month are based on 4-week intervals and are prorated to account for missing migraine reports. The number of migraine days per month were prorated to 28 days and derived for month (i.e., 4-week interval) in on-DBT efficacy analysis period as follows: 28*(total number of migraine days in month [Week 9 to 12])/ (total number of efficacy data days in month [Week 9 to 12])
Time Frame: Baseline, Week 9 to Week 12 of the DBT phase
Population: DBT migraine analysis set included participants in the DBT efficacy analysis set with >= 14 days of eDiary data (not necessarily consecutive) in both the OP and >= 1 month (4-week interval) during the DBT Phase.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rimegepant | Placebo
Number analyzed (Participants) | 240 | 244
Percentage of participants | 41.7 [35.5 to 47.9] | 34.4 [28.5 to 40.4]
Statistical Analysis 1: Comparison: Rimegepant vs Placebo; The percentages of participants with reductions were compared between treatment groups using Mantel-Haenszel risk estimation with stratification by randomization stratum (stable prophylactic migraine medication use throughout randomization; yes, no); Test type: Superiority; p = 0.0989, Mantel Haenszel — P-value >0.05; therefore, all secondary outcome measures listed after this outcome measure in the hierarchy were not tested; Difference in Percentage = 7.3, 95% CI 2-sided [-1.4 to 15.9]

3. Secondary Outcome: Mean Change From Baseline in Number of Migraine Days Per Month Over the Entire DBT Phase (Weeks 1 to 12)
Description: Migraine day:1) day of eDiary efficacy data with a qualified migraine headache, defined as: Headache lasted for >= 30 minutes and had 2 or more of following pain features: Unilateral and pulsating, moderate or severe pain intensity, worsen or avoid physical activity with one or more following associated symptoms: nausea, vomiting, both photophobia and phonophobia or 2) Acute migraine-specific medication day as eDiary efficacy data with a "yes" response to either of the 2 questions about taking triptan or ergotamine to treat headache or non-scheduled OL Rimegepant dosing day. In the model analysis, this outcome was also evaluated based on the monthly number of migraine days (and estimated the migraine days per month over the entire DBT phase). The number of migraine days per month were prorated to 28 days and derived for month (i.e.,4-week interval) in on-DBT efficacy analysis period as follows: 28*(total number of migraine days in month/ (total number of efficacy data days in month).
Time Frame: Baseline, Week 1 to Week 12 of the DBT phase
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Days/month
Arm/Group | Rimegepant | Placebo
Number analyzed (Participants) | 240 | 244
Days/month | -2.5 [-2.91 to -2.15] | -1.1 [-1.47 to -0.64]

4. Secondary Outcome: Mean Change From Baseline in Number of Migraine Days Per Month From Week 1 to 4 of the DBT Phase
Description: Migraine day: 1) day of eDiary efficacy data with a qualified migraine headache, defined as: Headache lasted for >= 30 minutes and had 2 or more of following pain features: Unilateral and pulsating, moderate or severe pain intensity, worsen or avoid physical activity with one or more of the following associated symptoms: nausea, vomiting, both photophobia and phonophobia or 2) Acute migraine-specific medication day as eDiary efficacy data with a "yes" response to either of the 2 questions about taking triptan or ergotamine to treat headache or non-scheduled OL Rimegepant dosing day. The number of migraine days per month were prorated to 28 days and derived for month (i.e., 4-week interval) in on-DBT efficacy analysis period as follows: 28*(total number of migraine days in month [Week 1 to 4])/ (total number of efficacy data days in month [Week 1 to 4]).
Time Frame: Baseline, Week 1 to Week 4 of the DBT phase
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Days/month
Arm/Group | Rimegepant | Placebo
Number analyzed (Participants) | 240 | 244
Days/month | -2.7 [-3.11 to -2.20] | -0.8 [-1.26 to -0.32]

5. Secondary Outcome: Mean Number of Acute Migraine-specific Medication Days Per Month From Week 9 to 12 of the DBT Phase
Description: An acute migraine-specific medication day was defined as day of eDiary efficacy data with a "yes" response to either of the 2 questions about taking triptan or ergotamine to treat headache or aura. Migraine days per month are assessed as "migraine days per 4 weeks" to correspond with the 4-week visit schedule. Migraine days per month are based on 4-week intervals and are prorated to account for missing migraine reports. The number of acute migraine-specific medication days per month was prorated to 28 days and derived for month (i.e., 4-week interval) in the on-DBT efficacy analysis period: 28*(total number of acute migraine-specific medication days in the month [Week 9 to 12])/ (total number of efficacy data days in the month [Week 9 to 12]).
Time Frame: Week 9 to Week 12 of the DBT phase
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Days/month
Arm/Group | Rimegepant | Placebo
Number analyzed (Participants) | 240 | 244
Days/month | 5.0 [4.40 to 5.55] | 5.8 [5.24 to 6.40]

6. Secondary Outcome: Mean Change From Baseline in the Migraine-Specific Quality-of-Life Questionnaire (MSQoL) v 2.1 Role Function - Restrictive Domain Score at Week 12 of the DBT Phase
Description: MSQoL is a self-administered, 14-item instrument validated in 3 domains: role restriction, role prevention, and the emotional function. The role function-restrictive domain consists of 7 items that describe how migraine limits one's daily social and work-related activities. Participants respond to items using a 6-point scale: "none of the time," "a little bit of the time," "some of the time," "a good bit of the time," "most of the time," and "all of the time," which are assigned scores of 1 to 6, respectively. Item scores are recoded using (7 - original score). Next, raw dimension scores are computed as a sum of recoded item scores and rescaled from a 0 to 100 scale such that higher scores indicate better quality of life. The change from baseline was calculated as the MSQoL restrictive role function domain score at Week 12 of the DBT phase minus the MSQoL restrictive role function domain score at baseline.
Time Frame: Baseline, Week 12 of the DBT phase
Population: DBT efficacy analysis set included participants in the full analysis set who (1) were randomized only once, and (2) took >= 1 dose of DB study intervention. Analysis was based on DBT efficacy analysis set with paired data (i.e., Non missing scores at both baseline and Week 12). Here, " Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Rimegepant | Placebo
Number analyzed (Participants) | 228 | 237
Score on a scale | 7.8 [6.20 to 9.44] | 3.7 [2.05 to 5.36]

7. Secondary Outcome: Mean Change From Baseline in the Migraine Disability Assessment Total Score (MIDAS) at Week 12 of the DBT Phase
Description: MIDAS is a retrospective, self-administered, 5-item questionnaire that measures headache-related disability as lost time due to headache from paid work or school, household work, and non-work activities. Participants provide the number of missed work or school days; missed household chores days; missed social or leisure activity days; and days at work or school, and separately at home, where productivity was reduced by half or more in the last 3 months (scale: 0 - 90 for each of 5 subscales). The 5 subscale scores are summed to compute the MIDAS total score (scale: 0 - 450). Lower scores indicate less headache-related disability. The change from baseline was calculated as the MIDAS total score at Week 12 of the DBT phase minus the MIDAS total score at baseline.
Time Frame: Baseline, Week 12 of the DBT phase
Population: DBT efficacy analysis set included participants in the full analysis set (FAS) who (1) were randomized only once, and (2) took >= 1 dose of DB study intervention. Analysis was based on DBT efficacy analysis set with paired data (i.e., Non missing scores at both baseline and Week 12). Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Rimegepant | Placebo
Number analyzed (Participants) | 228 | 237
Score on a scale | -4.0 [-5.57 to -2.42] | -1.6 [-3.88 to 0.70]

8. Secondary Outcome: Mean Change From Baseline in the EuroQol 5 Dimensions 5-level (EQ-5D-5L) Visual Analogue Scale (VAS) Score at Week 12 of the DBT Phase
Description: EQ-5D-5L is a standardized measure of health status. The EQ-5D-5L consisted of EQ-5D-5L descriptive system and the EQ VAS. For EQ VAS participant rated their overall health status from 0 (worst imaginable) to 100 (best imaginable), higher scores indicating a better health state.
Time Frame: Baseline, Week 12 of the DBT phase
Population: DBT efficacy analysis set included participants in the full analysis set who (1) were randomized only once, and (2) took >= 1 dose of DB study intervention. Analysis was based on DBT efficacy analysis set with paired data (i.e., nonmissing scores at both baseline and Week 12). Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Rimegepant | Placebo
Number analyzed (Participants) | 228 | 237
Score on a scale | 3.5 [1.60 to 5.37] | 0.8 [-1.40 to 3.02]

9. Secondary Outcome: Number of Participants With Adverse Events (AEs) By Intensity in DBT Phase
Description: An Adverse Event (AE) was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a participant or clinical investigation participant administered an investigational (medicinal) product and that does not necessarily have a causal relationship with this treatment. Definition of AE in terms of intensity: Mild: Is usually transient and may require only minimal treatment or therapeutic intervention. The event does not generally interfere with usual activities of daily living. Moderate: Is usually alleviated with additional specific therapeutic intervention. The event interferes with usual activities of daily living, causing discomfort but poses no significant or permanent risk of harm to the participant. Severe: Interrupts usual activities of daily living, significantly affects clinical status, or may require intensive therapeutic intervention.
Time Frame: From Day 1 of dosing up to 7 days post last dose of study drug in DBT phase or prior to start of OL rimegepant dose, whichever was earlier (maximum up to 13 weeks)
Population: Double-blind safety analysis set (DBSAS) included participants in the SAS who took >= 1 dose of DB study drug (Rimegepant or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant | Placebo
Number analyzed (Participants) | 247 | 249
Participants
  Any AE | 135 | 102
  Mild AE | 110 | 96
  Moderate AE | 24 | 6
  Severe AE | 1 | 0

10. Secondary Outcome: Number of Participants With AEs By Intensity in Open-Label Extension (OLE) Phase
Description: An AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a participant or clinical investigation participant administered an investigational (medicinal) product and that does not necessarily have a causal relationship with this treatment. Definition of AE in terms of intensity: Mild: Is usually transient and may require only minimal treatment or therapeutic intervention. The event does not generally interfere with usual activities of daily living. Moderate: Is usually alleviated with additional specific therapeutic intervention. The event interferes with usual activities of daily living, causing discomfort but poses no significant or permanent risk of harm to the participant. Severe: Interrupts usual activities of daily living, significantly affects clinical status, or may require intensive therapeutic intervention.
Time Frame: From Day 1 of OL Rimegepant dosing up to 7 days post last dose (maximum up to 41 weeks)
Population: Open label (OL) SAS included participants in the SAS who took >= 1 dose of OL Rimegepant.
Measure: Count of Participants; unit: Participants
Groups:
- DBT Rimegepant/OLE Rimegepant: Eligible participants continued to receive Rimegepant in a similar way from Week 12 to Week 52 (40 weeks) in the OLE period.
- DBT Placebo/OLE Rimegepant: Eligible participants continued to receive Rimegepant at a dose of 75 mg, orally as an ODT from Week 12 to Week 52 (40 weeks) in the OLE period.
Arm/Group | DBT Rimegepant/OLE Rimegepant | DBT Placebo/OLE Rimegepant
Number analyzed (Participants) | 227 | 231
Participants
  Any AE | 162 | 175
  Mild AE | 127 | 141
  Moderate AE | 33 | 33
  Severe AE | 2 | 1

11. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) in DBT Phase
Description: An AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a participant or clinical investigation participant administered an investigational (medicinal) product and that does not necessarily have a causal relationship with this treatment. A serious adverse event (SAE) was any untoward medical occurrence at any dose that: resulted in death; was life-threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/ incapacity; resulted in congenital anomaly/birth defect in the off spring who received rimegepant were considered an important medical event.
Time Frame: as for outcome 9
Population: DBSAS included participants in the SAS who took >= 1 dose of DB study drug (Rimegepant or placebo).
Measure: Count of Participants; unit: Participants
Groups:
- Rimegepant: Participants received Rimegepant at a dose of 75 mg, orally as an ODT, once EOD for 12 weeks in the DBT period.
Arm/Group | Rimegepant | Placebo
Number analyzed (Participants) | 247 | 249
Participants | 2 | 1

12. Secondary Outcome: Number of Participants With SAEs in OLE Phase
Description: An AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a participant or clinical investigation participant administered an investigational (medicinal) product and that does not necessarily have a causal relationship with this treatment. A SAE was any untoward medical occurrence at any dose that: resulted in death; was life-threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/ incapacity; resulted in congenital anomaly/birth defect in the offspring who received rimegepant were considered an important medical event.
Time Frame: From Day 1 of OL Rimegepant dosing up to 7 days post last dose (maximum up to 41 weeks)
Population: OLSAS included participants in the SAS who took >= 1 dose of OL Rimegepant.
Measure: Count of Participants; unit: Participants
Arm/Group | DBT Rimegepant/OLE Rimegepant | DBT Placebo/OLE Rimegepant
Number analyzed (Participants) | 227 | 231
Participants | 4 | 0

13. Secondary Outcome: Number of Participants With AEs Leading to Discontinuation of Study Drug in DBT Phase
Description: An AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a participant or clinical investigation participant administered an investigational (medicinal) product and that does not necessarily have a causal relationship with this treatment. In this outcome measure participants with adverse events leading to discontinuation of study drug were reported.
Time Frame: as for outcome 9
Population: DBSAS included participants in the SAS who took >= 1 dose of DB study drug (Rimegepant or placebo).
Measure: Count of Participants; unit: Participants
Groups:
- Rimegepant: Participants received RMG at a dose of 75 mg orally as an ODT, once EOD for 12 weeks in the DBT period.
Arm/Group | Rimegepant | Placebo
Number analyzed (Participants) | 247 | 249
Participants | 4 | 2

14. Secondary Outcome: Number of Participants With AEs Leading to Discontinuation of Study Drug in OLE Phase
Description: as for outcome 13
Time Frame: From Day 1 of OL Rimegepant dosing up at Week 12 to Week 52 (40 weeks)
Population: OLSAS included participants in the SAS who took >= 1 dose of OL Rimegepant.
Measure: Count of Participants; unit: Participants
Arm/Group | DBT Rimegepant/OLE Rimegepant | DBT Placebo/OLE Rimegepant
Number analyzed (Participants) | 227 | 231
Participants | 2 | 4

15. Secondary Outcome: Number of Participants With Grade 3 to 4 Laboratory Abnormalities in DBT Phase: Hematology Parameters
Description: The laboratory parameters were graded according to the National Cancer Institute (NCI) common terminology criteria for adverse events (CTCAE) version (v)5.0 severity grade. Grade 1=mild AE. Grade 2=moderate AE. Grade 3=severe AE and Grade 4=life-threatening consequences; urgent intervention indicated. Hematology parameters included: eosinophils, hemoglobin (high, low), lymphocytes (high, low), white blood cell count (WBC) (low, high), platelets, and neutrophils. hematocrit, red blood cell count, Number of participants with non-zero laboratory abnormalities of hematology parameters were reported in this outcome measure.
Time Frame: as for outcome 9
Population: DBSAS included participants in the SAS who took >= 1 dose of DB study drug (Rimegepant or placebo). Here, '' Overall Number of Participants Analyzed'' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant | Placebo
Number analyzed (Participants) | 241 | 243
Participants
  Hemoglobin, low | 2 | 0
  Neutrophils | 4 | 0
  Platelets | 1 | 0
  White blood cell count, low | 1 | 0

16. Secondary Outcome: Number of Participants With Grade 3 to 4 Laboratory Abnormalities in OLE Phase: Hematology Parameters
Description: The laboratory parameters were graded according to the NCI CTCAE v5.0 severity grade. Grade 1=mild AE. Grade 2=moderate AE. Grade 3=severe AE and Grade 4=life-threatening consequences; urgent intervention indicated. Hematology parameters included: eosinophils, hemoglobin (high, low), lymphocytes (high, low), WBC (low, high), platelets, and neutrophils. Number of participants with non-zero laboratory abnormalities of hematology parameters were reported in this outcome measure.
Time Frame: From Day 1 of OL Rimegepant dosing up to 7 days post last dose (maximum up to 41 weeks)
Population: OLSAS included participants in the SAS who took >= 1 dose of OL Rimegepant. Here, '' Overall Number of Participants Analyzed'' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | DBT Rimegepant/OLE Rimegepant | DBT Placebo/OLE Rimegepant
Number analyzed (Participants) | 226 | 231
Participants
  Hemoglobin, low | 2 | 1
  Lymphocytes, low | 1 | 1

17. Secondary Outcome: Number of Participants With Grade 3 to 4 Laboratory Abnormalities in DBT Phase: Serum Chemistry Parameters
Description: The laboratory parameters were graded according to the NCI CTCAE v5.0 severity grade. Grade 1=mild AE. Grade 2=moderate AE. Grade 3=severe AE. Grade 4=life-threatening consequences; urgent intervention indicated. Serum chemistry parameters included: creatine kinase, low density lipoprotein (LDL) cholesterol, LDL cholesterol, fasting, triglycerides, triglycerides, fasting and not fasting, alanine aminotransferase increased, albumin, alkaline phosphatase, aspartate aminotransferase increased, bicarbonate, bilirubin, calcium (high, low), cholesterol, creatinine, estimated glomerular filtration rate (eGFR), glucose (high, low), lactate dehydrogenase, LDL cholesterol, potassium (high, low), sodium (high, low), and uric acid. Number of participants with non-zero laboratory abnormalities of serum chemistry parameters were reported in this outcome measure.
Time Frame: as for outcome 9
Population: DBSAS included participants in the SAS who took >= 1 dose of DB study drug (Rimegepant or placebo). All participants reported under "Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row.
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant | Placebo
Number analyzed (Participants) | 247 | 249
Participants
  Creatine kinase: number analyzed (Participants) | 241 | 243
  Creatine kinase | 4 | 0
  LDL cholesterol: number analyzed (Participants) | 199 | 203
  LDL cholesterol | 0 | 4
  Triglycerides: number analyzed (Participants) | 199 | 204
  Triglycerides | 1 | 0

18. Secondary Outcome: Number of Participants With Grade 3 to 4 Laboratory Abnormalities in OLE Phase: Serum Chemistry Parameters
Description: The laboratory parameters were graded according to the NCI CTCAE v5.0 severity grade. Grade 1=mild AE. Grade 2=moderate AE. Grade 3=severe AE. Grade 4=life-threatening consequences; urgent intervention indicated. Serum chemistry parameters included: creatine kinase, LDL cholesterol, LDL cholesterol, triglycerides, triglycerides, alanine aminotransferase increased, albumin, alkaline phosphatase, aspartate aminotransferase increased, bicarbonate, bilirubin, calcium (high, low), cholesterol, creatinine, eGFR, glucose (high, low), lactate dehydrogenase, potassium (high, low), sodium (high, low), uric acid. Number of participants with non-zero laboratory abnormalities of serum chemistry parameters were reported in this outcome measure.
Time Frame: From Day 1 of OL Rimegepant dosing up to 7 days post last dose (maximum up to 41 weeks)
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | DBT Rimegepant/OLE Rimegepant | DBT Placebo/OLE Rimegepant
Number analyzed (Participants) | 225 | 231
Participants
  LDL cholesterol | 7 | 7
  Triglycerides | 1 | 1

19. Secondary Outcome: Number of Participants With Grade 3 to 4 Changes in DBT Phase: Urinalysis
Description: The laboratory parameters were graded according to the NCI CTCAE v5.0 severity grade. Grade 1=mild AE. Grade 2=moderate AE. Grade 3=severe AE and Grade 4=life-threatening consequences; urgent intervention indicated. Urinalysis parameters included: urine glucose and urine protein.
Time Frame: as for outcome 9
Population: DBSAS included participants in the SAS who took >= 1 dose of DB study drug (Rimegepant or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant | Placebo
Number analyzed (Participants) | 247 | 249
Participants | 0 | 0

20. Secondary Outcome: Number of Participants With Grade 3 to 4 Changes in OLE Phase: Urinalysis
Description: The laboratory parameters were graded according to the NCI CTCAE v5.0 severity grade. Grade 1=mild AE. Grade 2=moderate AE. Grade 3=severe AE and Grade 4=life-threatening consequences; urgent intervention indicated. Urinalysis parameters included: urine glucose and urine protein. Number of participants with non-zero laboratory abnormalities of urinalysis parameters were reported in this outcome measure.
Time Frame: From Day 1 of OL Rimegepant dosing up to 7 days post last dose (maximum up to 41 weeks)
Population: OLSAS included participants in the SAS who took >= 1 dose of OL Rimegepant. Here, ''Overall Number of Participants Analyzed'' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | DBT Rimegepant/OLE Rimegepant | DBT Placebo/OLE Rimegepant
Number analyzed (Participants) | 217 | 224
Participants | 3 | 1

21. Secondary Outcome: Number of Participants With Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) >3* Upper Lower Limit of Normal (ULN) Concurrent With Total Bilirubin (TBIL) >2*ULN in DBT Phase
Description: Number of participants with ALT or AST >3*ULN concurrent with TBIL >2*ULN in DBT phase were reported in this outcome measure.
Time Frame: as for outcome 9
Population: DBSAS included participants in the SAS who took >= 1 dose of DB study drug (Rimegepant or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant | Placebo
Number analyzed (Participants) | 247 | 249
Participants | 0 | 0

22. Secondary Outcome: Number of Participants With ALT or AST> 3* ULN Concurrent With TBIL >2* ULN in OLE Phase
Description: Number of participants with ALT or AST >3*ULN concurrent with TBIL >2*ULN in OLE phase were reported in this outcome measure.
Time Frame: From Day 1 of OL Rimegepant dosing up to 7 days post last dose (maximum up to 41 weeks)
Population: OLSAS included participants in the SAS who took >= 1 dose of OL Rimegepant.
Measure: Count of Participants; unit: Participants
Arm/Group | DBT Rimegepant/OLE Rimegepant | DBT Placebo/OLE Rimegepant
Number analyzed (Participants) | 227 | 231
Participants | 0 | 0

23. Secondary Outcome: Number of Participants With Hepatic-related AEs in the DBT Phase
Description: An AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a participant or clinical investigation participant administered an investigational (medicinal) product and that does not necessarily have a causal relationship with this treatment. Hepatic AEs included cirrhosis, hepatic failure, hepatitis, jaundice, or liver failure.
Time Frame: as for outcome 9
Population: DBSAS included participants in the SAS who took >= 1 dose of DB study drug (Rimegepant or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant | Placebo
Number analyzed (Participants) | 247 | 249
Participants | 3 | 4

24. Secondary Outcome: Number of Participants With Hepatic-related AEs in the OLE Phase
Description: as for outcome 23
Time Frame: From Day 1 of OL Rimegepant dosing up to 7 days post last dose (maximum up to 41 weeks)
Population: OLSAS included participants in the SAS who took >= 1 dose of OL Rimegepant.
Measure: Count of Participants; unit: Participants
Arm/Group | DBT Rimegepant/OLE Rimegepant | DBT Placebo/OLE Rimegepant
Number analyzed (Participants) | 227 | 231
Participants | 8 | 7

25. Secondary Outcome: Number of Participants With Hepatic-related AEs Leading to Study Drug Discontinuation in the DBT Phase
Description: An AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a participant or clinical investigation participant administered an investigational (medicinal) product and that does not necessarily have a causal relationship with this treatment. Hepatic AEs included cirrhosis, hepatic failure, hepatitis, jaundice, or liver failure. Number of participants with Hepatic-related AEs leading to study drug discontinuation were reported in this outcome measure.
Time Frame: as for outcome 9
Population: DBSAS included participants in the SAS who took >= 1 dose of DB study drug (Rimegepant or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant | Placebo
Number analyzed (Participants) | 247 | 249
Participants | 0 | 1

26. Secondary Outcome: Number of Participants With Hepatic-related AEs Leading to Study Drug Discontinuation in the OLE Phase
Description: as for outcome 25
Time Frame: From Day 1 of OL Rimegepant dosing up to 7 days post last dose (maximum up to 41 weeks)
Population: OLSAS included participants in the SAS who took >= 1 dose of OL Rimegepant.
Measure: Count of Participants; unit: Participants
Arm/Group | DBT Rimegepant/OLE Rimegepant | DBT Placebo/OLE Rimegepant
Number analyzed (Participants) | 227 | 231
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: DBT phase: From Day 1 of dosing up to 7 days post last dose of study drug in DBT phase or prior to start of OL rimegepant dose, whichever was earlier (maximum up to 13 weeks); OLE phase: From Day 1 of OL Rimegepant dosing up to 7 days post last dose (maximum up to 41 weeks)
Description: Same event may appear as AE & serious adverse events (SAE), what is presented are distinct events. Event may be categorized as serious in 1 and as non-SAE in another participant, or 1 participant may have experienced both serious & non-SAE. DBSAS included participants in the SAS who took >= 1 dose of DB study drug (Rimegepant or placebo). OLSAS included participants in the SAS who took >= 1 dose of OL Rimegepant. For DBT phase MedDRA version v26.1 and for OLE phase version 27.1 was used.
Groups:
- DBT: Rimegepant: Participants received Rimegepant at a dose of 75 mg, orally as an ODT, once EOD for 12 weeks in the DBT period. Eligible participants continued to receive Rimegepant in a similar way from Week 12 to Week 52 (40 weeks) in the OLE period.
- DBT: Placebo: Participants received placebo, orally as an ODT, once EOD for 12 weeks in the DBT period. Eligible participants continued to receive Rimegepant at a dose of 75 mg, orally as an ODT from Week 12 to Week 52 (40 weeks) in the OLE period.
Arm/Group | DBT: Rimegepant | DBT: Placebo | DBT Rimegepant/OLE Rimegepant | DBT Placebo/OLE Rimegepant
All-Cause Mortality (participants affected / at risk) | 0/247 | 0/249 | 0/227 | 0/231
Serious Adverse Events (participants affected / at risk) | 2/247 | 1/249 | 4/227 | 0/231
Other Adverse Events (participants affected / at risk) | 85/247 | 73/249 | 148/227 | 150/231
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DBT: Rimegepant (N=247) | DBT: Placebo (N=249) | DBT Rimegepant/OLE Rimegepant (N=227) | DBT Placebo/OLE Rimegepant (N=231)
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Nodal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Coronavirus infection (Infections and infestations) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DBT: Rimegepant (N=247) | DBT: Placebo (N=249) | DBT Rimegepant/OLE Rimegepant (N=227) | DBT Placebo/OLE Rimegepant (N=231)
Abdominal discomfort (Gastrointestinal disorders) | 3 | 3 | 1 | 4
Abdominal pain upper (Gastrointestinal disorders) | 8 | 2 | 7 | 8
Constipation (Gastrointestinal disorders) | 7 | 1 | 8 | 8
Dental caries (Gastrointestinal disorders) | 1 | 3 | 8 | 4
Diarrhoea (Gastrointestinal disorders) | 3 | 4 | 6 | 4
Nausea (Gastrointestinal disorders) | 3 | 4 | 0 | 0
Toothache (Gastrointestinal disorders) | 3 | 2 | 8 | 5
Pyrexia (General disorders) | 6 | 5 | 7 | 12
Bronchitis (Infections and infestations) | 1 | 3 | 4 | 4
COVID-19 (Infections and infestations) | 6 | 7 | 32 | 28
Coronavirus infection (Infections and infestations) | 8 | 4 | 12 | 10
Influenza (Infections and infestations) | 5 | 5 | 11 | 14
Nasopharyngitis (Infections and infestations) | 21 | 25 | 51 | 64
Pharyngitis (Infections and infestations) | 3 | 1 | 5 | 3
Sinusitis (Infections and infestations) | 3 | 0 | 7 | 6
Blood creatine phosphokinase increased (Investigations) | 3 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 6 | 15 | 9
Dysmenorrhoea (Reproductive system and breast disorders) | 3 | 0 | 3 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 8 | 11 | 10
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 3 | 3 | 4
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 6 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 3 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 2 | 4
Dry eye (Eye disorders) | 0 | 0 | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 6 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 3 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 6 | 3
Fatigue (General disorders) | 0 | 0 | 4 | 0
Cystitis (Infections and infestations) | 0 | 0 | 4 | 5
Gastroenteritis (Infections and infestations) | 0 | 0 | 6 | 7
Oral herpes (Infections and infestations) | 0 | 0 | 3 | 3
Heat illness (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 4
Medication error (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 4
Dizziness (Nervous system disorders) | 0 | 0 | 3 | 3
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 3
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 4 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 6
Hypertension (Vascular disorders) | 0 | 0 | 1 | 4
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 4 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 3 | 2
Enteritis infectious (Infections and infestations) | 0 | 0 | 0 | 3
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 3
Tonsillitis (Infections and infestations) | 0 | 0 | 3 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 4 | 3
Alanine aminotransferase increased (Investigations) | 0 | 0 | 4 | 5
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 3
Liver function test increased (Investigations) | 0 | 0 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 7 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 3
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-08-04): https://cdn.clinicaltrials.gov/large-docs/85/NCT05399485/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-23): https://cdn.clinicaltrials.gov/large-docs/85/NCT05399485/SAP_001.pdf